CLINICAL TRIAL: NCT01704183
Title: Effect of Fingolimod on the Cardiac Autonomic Regulation in Patients With Multiple Sclerosis
Acronym: FingoHRV
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2012-SS; 2012-002694-66 (EudraCT Number)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Relapse-remitting Multiple Sclerosis
Keywords: relapse-remitting multiple sclerosis; heart rate variability; fingolimod; cardiac autonomic regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to study the effect of fingolimod on cardiac autonomic regulation in patients with relapse-remitting multiple sclerosis.

This will be done by measuring heart rate variability from the 24-hour Holter recording and myocardial ventricular repolarisation patterns from the 12-lead electrocardiogram tracings.

The fingolimod treatment is prescribed according to the accepted drug label.

DETAILED DESCRIPTION:
The study will include 30 relapse-remitting multiple sclerosis patients. Assessments of heart rate variability and myocardial ventricular repolarisation pattern will be done 1) before fingolimod, 2) first day of fingolimod 3) after 3 months use and 4) after 12 months use of fingolimod.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years
* Understands the proposed research and actions to be taken
* The written informed consent has given
* clinical indication to fingolimod-treatment

Exclusion Criteria:

* Patient refuses
* Patient takes or has taken part in other clinical drug trial during the last month
* No clinical indication to the use of fingolimod
* Contraindication to the use of fingolimod

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurological clinic
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
change in heart rate variability | prior medication vs initiation vs 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Sakari Simula, MD, PhD, Study Director — Mikkeli Central Hospital, Department of Neurology; Päivi Hartikainen, MD, PhD, Study Director — Kuopio University Hospital, Neuro Center; Juha Hartikainen, MD, PhD, Study Director — Kuopio University Hospital, Heart Center
Locations (2):
- Finland (2):
  - Neuro Center, Kuopio University Hospital, Kuopio
  - Department of Neurology, Mikkeli Central Hospital, Mikkeli

REFERENCES:
- [Derived] Simula S, Laitinen TP, Laitinen TM, Hartikainen P, Hartikainen JE. Heart rate variability predicts the magnitude of heart rate decrease after fingolimod initiation. Mult Scler Relat Disord. 2016 Nov;10:86-89. doi: 10.1016/j.msard.2016.09.012. Epub 2016 Sep 30. PMID 27919506
- [Derived] Simula S, Laitinen T, Laitinen TM, Tarkiainen T, Hartikainen P, Hartikainen JE. Effect of fingolimod on cardiac autonomic regulation in patients with multiple sclerosis. Mult Scler. 2016 Jul;22(8):1080-5. doi: 10.1177/1352458515604384. Epub 2015 Sep 11. PMID 26362903
- [Derived] Simula S, Laitinen T, Laitinen TM, Tarkiainen T, Hartikainen JE, Hartikainen P. Effects of Three Months Fingolimod Therapy on Heart Rate. J Neuroimmune Pharmacol. 2015 Dec;10(4):651-4. doi: 10.1007/s11481-015-9619-8. Epub 2015 Jun 20. PMID 26092537